CLINICAL TRIAL: NCT00348686
Title: A Multicenter, Non-comparative, Phase IV Study to Evaluate the Effect of Candesartan Based Therapy in the Percent Change of proBNP Level After 24 Week Treatment in the Patients With Hypertension With Left Ventricular Hypertrophy
Brief Title: Candesartan Effectiveness Study in Pro-B Type Natriuretic Peptides (BNP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2452L00012; CAP
Record Dates: First submitted 2006-07-03; First posted 2006-07-06 (Estimated); Results first posted 2012-04-02 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Hypertension; Left Ventricular Hypertrophy
Keywords: LVH
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — candesartan; candesartan cilexetil; Felodipine

ARMS (1):
- Candesartan (Experimental): Subjects were treated for 24 weeks with Candesartan 16mg once daily as initial dose. Subjects were modified investigational product dose to Candesartan 32mg, Candesartan 32mg + Felodipine 5mg, Candesartan 32mg + Felodipine 10mg, sequentially according to their blood pressures.
  Interventions: Drug: Candesartan; Drug: Felodipine

INTERVENTIONS:
Drug: Candesartan — 16 mg once daily in oral tablet form
  Other Names: Atacand
Drug: Candesartan — 32 mg once daily in oral tablet form
  Other Names: Antacand
Drug: Felodipine — 5 mg once daily in oral tablet form
Drug: Felodipine — 10 mg once daily in oral tablet form

SUMMARY:
The purpose of this study is to investigate effect of candesartan based therapy on percent change of B type natriuretic peptides(BNP) level in the subjects with hypertension and left ventricular hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension with diastolic blood pressure within 95-115 mm/Hg or/and systolic blood pressure within 160-200 mm/Hg
* Patients diagnosed as left ventricular hypertrophy by electrocardiogram

Exclusion Criteria:

* Secondary hypertension
* History of myocardial infarction
* Stroke within the previous 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JeeWoong Son, MD, Study Director — AstraZeneca
Locations (11):
- South Korea (11):
  - Research Site, Busan
  - Research Site, Cheonan
  - Research Site, Cheongju-si
  - Research Site, Chunbuk
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gyungsangnamdo
  - Research Site, Jeonju
  - Research Site, Kwangju
  - Research Site, Pusan
  - Research Site, Ulsan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Milestone date: 15 June 2006 (FSI) ~ 05 June 2008 (LSLV) Type of location: General Hospital; 333 subjects enrolled, but 18 subjects failed to be randomized, 315 subjects were randomized to study.
Pre-assignment Details: Screening period: Laboratory test (Creatinine, potassium, ALT, etc)
Period: Overall Study
Arm/Group | Candesartan
Started | 315
Completed | 249
Not Completed | 66
Not completed — Withdrawal by Subject | 45
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 6
Not completed — Lost to Follow-up | 2
Not completed — Multiple Reasons | 8

BASELINE CHARACTERISTICS:
Arm/Group | Candesartan
Number analyzed (Participants) | 315
Age Continuous [Mean (Standard Deviation); unit: years]
  Average age of subjects who participated | 49.90 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 234

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of B Type Natriuretic Peptides (BNP) Level
Description: Change of B Type Natriuretic Peptides Level of the Subjects With Hypertension and Left Ventricular Hypertrophy (LVH) Treated With Candesartan Based Therapy for 24 Weeks was calculated just as the later time point minus the earlier time point. No specific calculation was used.
Time Frame: At Baseline and 24 weeks
Population: Followed Intent-to-treat analysis
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Candesartan
Number analyzed (Participants) | 292
Percent Change | -29.2 [-35.3 to -16.7]

2. Secondary Outcome: LVH(Left Ventricular Hypertrophy) Regression by Echocardiac Parameter, Left Ventricular Mass Index
Description: Change of Left Ventricular Hypertrophy(LVH) by Echocardiac Parameter, Left Ventricular mass Index (LVMI) was calculated and collected through the way of Last Observational carried forward. LVH/Index was calculated like this: Divide LV mass with Body Surface Area.
Time Frame: At Baseline and 24 weeks
Population: Only 245 patients who have reliable Echocardiac data were analyzed.
Measure: Median (Full Range); unit: g/m^2
Arm/Group | Candesartan
Number analyzed (Participants) | 245
g/m^2 | -10.90 [-14.00 to -7.0]

3. Secondary Outcome: Change of Systolic Blood Pressure (SBP)
Description: Change of Systolic Blood Pressure was calculated and collected through the way of Last Observational carried forward.
Time Frame: At Baseline and 24 weeks
Population: Only who has systolic blood pressure data both baseline and follow up was analyzed. Most of patient who enrolled, 302 have a data.
Measure: Median (Full Range); unit: mmHg
Arm/Group | Candesartan
Number analyzed (Participants) | 302
mmHg | -32.0 [-35.0 to -30.0]

4. Secondary Outcome: Change of Diastolic Blood Pressure (DBP)
Description: Change of Diastolic Blood Pressure was calculated and collected through the way of Last Observational carried forward.
  Only who has diastolic blood pressure data both baseline and follow up was analyzed. Most of patient who enrolled, 302 have a data.
Time Frame: At Baseline and 24 weeks
Population: Last Observational carried forward
Measure: Median (Full Range); unit: mmHg
Arm/Group | Candesartan
Number analyzed (Participants) | 302
mmHg | -20.0 [-20.0 to -18.0]

5. Secondary Outcome: Percent Change of proBNP(B Type Natriuretic Peptides) in Patients Treated With Candesartan Only
Description: Percent change of proBNP(B type Natriuretic Peptides) was calculated and collected through the way of Last Observational carried forward.
Time Frame: At Baseline and 24 weeks
Population: Only 201 patients are available for analysis.
Measure: Median (Full Range); unit: percent change
Arm/Group | Candesartan
Number analyzed (Participants) | 201
percent change | -18.9 [-33.0 to -6.6]

6. Secondary Outcome: Percent Change of proBNP(B Type Natriuretic Peptides) in Patients With Candesartan Plus Felodipine
Description: as for outcome 5
Time Frame: At Baseline and 24 weeks
Population: Only 91 patients are available for analysis
Measure: Median (Full Range); unit: percent change
Arm/Group | Candesartan
Number analyzed (Participants) | 91
percent change | -36.1 [-57.9 to -24.3]

ADVERSE EVENTS:
Arm/Group | Candesartan
Serious Adverse Events (participants affected / at risk) | 8
Other Adverse Events (participants affected / at risk) | 37
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Candesartan
Left paraduodenal hernia (Gastrointestinal disorders) | 1/315
Rectal prolapse aggravated (Gastrointestinal disorders) | 1/315
Cerebral infarction (Vascular disorders) | 1/315
Uterine myoma aggravated (Renal and urinary disorders) | 1/315
Cervical disc herniation aggravated (General disorders) | 1/315
Pneumonia with effusion in the right chest (Respiratory, thoracic and mediastinal disorders) | 1/315
Granuloma inguinale (Skin and subcutaneous tissue disorders) | 1/315
Acute myocardial infarction (Cardiac disorders) | 1/315
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Candesartan
Headache (Nervous system disorders) | 23/315
Dizziness (Nervous system disorders) | 16/315

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less